CLINICAL TRIAL: NCT03565406
Title: A Phase 1b Study of the Selective HDAC Inhibitor Mocetinostat in Combination With Ipilimumab and Nivolumab in Patients With Unresectable Stage III or Stage IV Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: recruiting or enrolling participants has halted prematurely and will not resume; participants are no longer being examined or treated
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00861
Record Dates: First submitted 2018-06-12; First posted 2018-06-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Unresectable Stage III or Stage IV Melanoma (Experimental)
  Interventions: Drug: Mocetinostat Induction Phase + Ipilimumab + Nivolumab; Drug: Mocetinostat Maintenance Phase + Ipilimumab + Nivolumab

INTERVENTIONS:
Drug: Mocetinostat Induction Phase + Ipilimumab + Nivolumab — Treatment Cycle 1: Mocetinostat at a dose of 90 mg PO TIW; ipilimumab will be administered IV at a dose of 1 mg/kg and nivolumab will be administered IV at a dose of 3 mg/kg during the 12-week induction period. The induction phase will last for 2 treatment cycles.
  Treatment Cycle 2: Mocetinostat at a dose of 70 mg PO TIW ipilimumab will be administered IV at a dose of 1 mg/kg and nivolumab will be administered IV at a dose of 3 mg/kg during the 12-week induction period. The induction phase will last for 2 treatment cycles.
Drug: Mocetinostat Maintenance Phase + Ipilimumab + Nivolumab — De-escalation Phase 1: Mocetinostat will be administered 50 mg PO TIW during each 84-day treatment cycle. Ipilimumab will be administered IV at a dose of 1 mg/kg and nivolumab will be administered IV at a dose of 3 mg/kg
  De-escalation Maintenance Phase 2: Mocetinostat will be administered 40 mg PO TIW during each 84-day treatment cycle. Ipilimumab will be administered IV at a dose of 0.3 mg/kg and nivolumab will be administered IV at a dose of 1 mg/kg during period

SUMMARY:
This is a Phase 1b, open-label, dose-escalation cohort study. The study will consist of a dose escalation assessment of the safety and tolerability of Mocetinostat administered concurrently in combination with ipilimumab and nivolumab to patients with advanced melanoma. Treatment will be divided into induction and maintenance phases. It is anticipated that this clinical study will enable selection of the RP2D and dose schedule of this 3-drug combination for further clinical testing. The trial will include an assessment of the pharmacodynamic activity of Mocetinostat administered in combination with ipilimumab and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed and dated an Institutional Review Board/Independent Ethics Committee -approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
* All patients must be either Stage IIIb/c or Stage IV according to the American Joint Committee on Cancer (AJCC) (7th edition) and have histologically-confirmed melanoma that is felt to be surgically unresectable in order to be eligible. Please refer to the AJCC Cancer Staging Manual, 7th edition for a description of tumor, lymph node, metastasis and staging.
* All melanomas, except ocular/uveal melanoma, regardless of primary site of disease will be allowed; mucosal melanomas are eligible.
* Patients must not have received prior anticancer treatment for metastatic disease (for example, but not limited to, systemic, local, radiation, radiopharmaceutical).
* Exceptions: Surgery for melanoma and/or postresection brain radiotherapy (RT) if central nervous system (CNS) metastases and/or prior treatment with adjuvant interferon (IFN) (as described in Exclusion Criterion 2).

  --All patients must have their disease status documented by a complete physical examination and imaging studies within 4 weeks prior to the first dose of study drug. Imaging studies must include computerized tomography (CT) scan of neck, chest, abdomen, pelvis, and all known sites of resected disease in the setting of Stage IIIb/c or Stage IV disease, and brain magnetic resonance imaging ([MRI], brain CT allowable if MRI is contraindicated).
* The complete set of baseline radiographic images must be available before treatment initiation.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Tumor tissue from the resected site of disease must be provided for biomarker analyses
* Prior treated CNS metastases must be without MRI evidence of recurrence for at least 4 weeks after treatment. Patients must be off immunosuppressive doses of systemic steroids (≥ 10 mg/day prednisone or equivalent) for at least 14 days prior to study drug administration, and must have returned to neurologic baseline status postoperatively

  * The 4-week period of stability is measured after the completion of the neurologic interventions (ie, surgery and/or radiation).
* In addition to neurosurgery to treat CNS metastases, adjuvant radiation after the resection of CNS metastasis is allowed. Immunosuppressive doses of systemic steroids (doses ≥ 10 mg/day prednisone or equivalent) must be discontinued at least 14 days before study drug administration.
* Prior surgery that required general anesthesia must be completed at least 4 weeks before study drug administration. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration.
* All baseline laboratory requirements will be assessed and should be obtained within 14 days of first dose of study drug. Screening laboratory values must meet the following criteria:
* White blood cells ≥ 2000/µL
* Neutrophils ≥ 1500/µL
* Platelets ≥ 100 × 10³/µL
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance > 40 mL/minute (using Cockcroft/Gault formula)
* Patient Re-enrollment: This study permits the re-enrollment of a patient that has discontinued the study as a screen failure (ie, patient has not been dosed/has not been treated). If re-enrolled, the patient must be re-consented.
* Males and females ≥ 18 years of age.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin hormone) within 24 hours prior to the start of study drug.; Women must not be breastfeeding.
* Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug plus 30 days (duration of ovulatory cycle). The half-lives of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. Given the blinded nature of this study, WOCBP should therefore use an adequate method to avoid pregnancy for a total of 23 weeks posttreatment completion.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half lives of the study drug(s) plus 90 days (duration of sperm turnover). The half-lives of nivolumab and ipilimumab are up to 25 days and 18 days, respectively. Given the blinded nature of this study, men should therefore use an adequate method of contraception for a total of 31 weeks posttreatment completion.
* Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section.

Exclusion Criteria:

* Patients with carcinomatosis meningitis or a history of ocular/uveal melanoma are excluded.
* Patients with previous nonmelanoma malignancies are excluded unless a complete resection or remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period (exceptions include, but are not limited to, nonmelanoma skin cancers, in situ bladder cancer, in situ gastric cancer or gastrointestinal stromal tumor, in situ colon cancers, in situ cervical cancers/dysplasia, or breast carcinoma in situ).
* Patients with active, known, or suspected autoimmune disease. Patients with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the Principal Investigator be consulted prior to signing informed consent.
* Patients with a condition requiring systemic treatment with either corticosteroids (≥ 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
* Prior therapy for melanoma with the following exceptions which are allowed: 1) surgery for the melanoma lesion(s), 2) adjuvant RT after neurosurgical resection for CNS lesions, and 3) prior adjuvant IFN (see qualifier below). Specifically, patients who received prior therapy with anti-PD-1, anti PD L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T cell costimulation or checkpoint pathways) are not eligible. • Prior treatment with adjuvant IFN is allowed if completed ≥ 3 months prior to treatment.
* Treatment directed against the melanoma (eg, chemotherapy, targeted agents, biotherapy, limb perfusion) that is administered after a prior complete resection other than adjuvant radiation after neurosurgical resection and IFN for resected melanoma.
* Previous therapy with histone deacetylase inhibitor.
* Any of the following laboratory abnormalities:
* ANC < 1,500/µL
* Platelet count < 100,000/µL
* Hematologic growth factors are not allowed at screening or during the first cycle of treatment
* Hemoglobin < 9 g/dL (< 5.5 mmol/L; previous red blood cell transfusion is permitted)
* Creatinine > 1.5 × ULN
* AST or ALT > 2.5 × ULN. For patients with liver metastasis, AST or ALT > 5 × ULN
* Serum total bilirubin > 1.5 mg/dL or > 3 × ULN for patients with hereditary benign hyperbilirubinemia
* Corrected QT interval (QTc) using Fridericia's formula value > 480 msec at screening; family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy at screening; previous history of drug induced QTc prolongation or the need for treatment with medications known or suspected of producing prolonged QTc intervals on electrocardiogram (ECG).
* Congestive heart failure (New York Heart Association Class III or IV), myocardial infarction within 12 months before starting study treatment, or unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris.
* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the Investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patient to receive protocol therapy.
* Any positive test result for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
* Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome.
* History of Grade ≥ 3 allergy to human monoclonal antibodies.
* Prisoners or patients who are involuntarily incarcerated.
* Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
* Pregnant or nursing women.
* Psychological, familial, sociological, or geographical conditions that potentially hamper compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Number of Dose Limiting Toxicities (DLTs), defining the maximum tolerated dose (MTD) | 60 Months

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of Mocetinostat administered in combination with ipilimumab and nivolumab | 60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weber, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Weber JS, Levinson BA, Laino AS, Pavlick AC, Woods DM. Clinical and immune correlate results from a phase 1b study of the histone deacetylase inhibitor mocetinostat with ipilimumab and nivolumab in unresectable stage III/IV melanoma. Melanoma Res. 2022 Oct 1;32(5):324-333. doi: 10.1097/CMR.0000000000000818. Epub 2022 Jun 9. PMID 35678233